CLINICAL TRIAL: NCT03937817
Title: Collection of Human Biospecimens for Basic and Clinical Research Into Globin Variants
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190093; 19-I-0093
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09-17

CONDITIONS: Alpha and Beta Thalassemia; Sickle Cell Disease; Malaria; Human Physiology
Keywords: Assay Development; Malaria; Sickle Cell Disease; Alpha and Beta Thalassemia; Natural History
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell; Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy volunteers and patients with hematologic and hemolytic diseases, including alpha and beta globin variants, sickle cell disease, malaria, or other diseases involving inflammation or endothelial dysfunction.

SUMMARY:
Background:

Blood disorders like sickle cell disease and malaria affect many people around the world. Researchers want to learn more about blood disorders. To do this, they need to collect biological samples from people with blood disorders. They also need to collect samples from healthy people.

Objective:

To collect samples to use for research on blood disorders.

Eligibility:

People ages 18-70 who have blood disorders. Healthy volunteers without blood disorders are also needed.

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests.

Participants will give one or more samples. They will give them over 5 years. They can choose not to give any of the samples:

Saliva: Participants will spit into a tube. They may also have the inside of their mouth swabbed.

Urine: Participants will urinate into a cup.

Blood and blood waste products: Blood will be taken through a needle in the participant s arm.

Fat samples: An area on the participant s belly or buttock will be numbed. A small cut will be made into the skin and a small piece of fat removed.

Mucus and cells from the lungs: The participant will be sedated. A flexible tube will be inserted through the nose or mouth into the lung airways. These participants will also have a physical exam, chest x-ray, and heart tests after the procedure.

DETAILED DESCRIPTION:
The Physiology Unit of the Laboratory of Malaria and Vector Research studies the role of globin variants in erythroid and non-erythroid tissues. We hope to better understand the mechanism(s) through which alpha and beta globin variants impact malaria, sickle cell disease, or other diseases involving inflammation or vascular endothelial dysfunction.

The collection of human specimens from healthy volunteers and patients with malaria, sickle cell disease, or other diseases involving inflammation or endothelial dysfunction is necessary for the development of laboratory and physiological assays to further basic and clinical research studies. This protocol defines the purposes for which specimens will be collected and establishes general conditions under which sample collection will be performed. Development of assays and our research into the roles of alpha and beta globin in normal human physiology, as well as in the pathogenesis of malaria and sickle cell disease, requires laboratory analysis of saliva/buccal swab, urine, blood, blood waste products, adipose tissue, bronchial brushing, and/or bronchoalveolar lavage specimens from human volunteers.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

  1. Aged 18-70 years.
  2. Able to provide informed consent.
  3. Willing to allow biological samples to be stored for future research.
  4. Willing to provide one or more of the following tissues: saliva, urine, blood, blood waste products, adipose tissue, bronchial brushing, and/or BAL samples.
  5. Willing to allow genetic testing on collected biological samples.

     PARTICIPANT EXCLUSION CRITERIA:
* Exclusion Criteria for All Participants

The following exclusion criteria apply to all participants who will provide any of the following samples in-person at the NIH CC: saliva, urine, blood, blood waste products, adipose tissue, bronchial brushing, and/or BAL samples:

1. Pregnancy.
2. Positive testing for hepatitis B virus, hepatitis C virus, or HIV (as determined by serum screening tests or relevant viral quantitative studies.)
3. Any condition that requires active medical intervention or monitoring to avert serious danger to the individual s health or wellbeing.
4. Any condition that, in the opinion of the PI, contraindicates participation in this study.

   * Additional Exclusion Criteria for Individuals Giving Blood for Research

1. Hemoglobin < 10 g/dL for healthy female volunteers, < 12 g/dL for healthy male volunteers, or < 6 g/dL for participants with sickle cell disease or other chronic anemias.

-Additional Exclusion Criteria for Adipose Tissue Biopsy

Individuals meeting any of the following criteria will be excluded from undergoing adipose tissue biopsy. If the participant no longer meets any of these criteria at a later time, then they will be allowed to undergo this procedure.

1. Currently taking anticoagulation medication.
2. Platelets < 100,000/microL.
3. History of keloid formation (or irregular fibrous tissue formed at the site of a scar or injury).
4. History of adverse reactions to lidocaine or other local anesthetics.
5. Any condition that, in the opinion of the PI, contraindicates this procedure.

Use of aspirin (or acetylsalicylic acid) and nonsteroidal anti-inflammatory drugs (NSAIDs) are permitted.

-Additional Exclusion Criteria for Bronchoscopy

Individuals meeting any of the following criteria will be excluded from undergoing bronchoscopy. If the participant no longer meets any of these criteria at a later time, then they will be allowed to undergo this procedure.

1. Prothrombin time (PT) > 1 second above the upper limit of normal (ULN) or international normalized ratio > 1.3.
2. Partial thromboplastin time (PTT) > 1 second above ULN.
3. Platelets < 150,000/microL.
4. Currently taking anticoagulation medication.
5. Use of aspirin within 2 weeks of the bronchoscopy or NSAIDs within 2 days of the bronchoscopy.
6. Diagnosis of a pulmonary disorder (eg, asthma, chronic bronchitis, cystic fibrosis, or bronchiectasis).
7. Respiratory tract infection within the last 4 weeks.
8. History of adverse reactions to systemic and/or local anesthetics that will be used for this procedure.
9. History of cigarette smoking within the past 3 months.
10. History of chronic opioid use.
11. History of drug or alcohol abuse.
12. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 40% of predicted or pre-bronchodilator FEV1 < 35% of predicted.
13. Active bronchospasm on physical examination.
14. History of lidocaine allergy.
15. Any condition that, in the opinion of the PI, contraindicates this procedure.

Co-enrollment guidelines: Participants may be co-enrolled in other studies. However, the PI must be notified of co-enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants may be recruited from other NIH protocols, the NIH Clinical Research Healthy Volunteer Program, patient recruitment websites for the National Heart, Lung, and Blood Institute, community outreach, ResearchMatch, and clinicaltrials.gov.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Collect biological specimens (saliva, urine, blood, blood waste products, adipose tissue, bronchial brushing, and/or BAL) | Throughout study
  Development and optimization of scientific assays and research of globin variants, sickle cell disease, malaria, or other related diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Ackerman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This protocol is not a clinical trial and has no intervention. We do not currently have a plan to share individual participant data (IPD). The IRB-approved data sharing plan in our protocol is as follows: "Identified human data generated in this study will be shared for future research in the Biomedical Translational Research Information System (automatic for activities in the CC). De-identified data may also be shared with outside collaborators under appropriate agreements."

REFERENCES:
- [Background] Embury SH, Dozy AM, Miller J, Davis JR Jr, Kleman KM, Preisler H, Vichinsky E, Lande WN, Lubin BH, Kan YW, Mentzer WC. Concurrent sickle-cell anemia and alpha-thalassemia: effect on severity of anemia. N Engl J Med. 1982 Feb 4;306(5):270-4. doi: 10.1056/NEJM198202043060504. PMID 6172710
- [Background] Piel FB, Weatherall DJ. The alpha-thalassemias. N Engl J Med. 2014 Nov 13;371(20):1908-16. doi: 10.1056/NEJMra1404415. PMID 25390741
- [Background] Straub AC, Lohman AW, Billaud M, Johnstone SR, Dwyer ST, Lee MY, Bortz PS, Best AK, Columbus L, Gaston B, Isakson BE. Endothelial cell expression of haemoglobin alpha regulates nitric oxide signalling. Nature. 2012 Nov 15;491(7424):473-7. doi: 10.1038/nature11626. Epub 2012 Oct 31. PMID 23123858
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0093.html